CLINICAL TRIAL: NCT03587649
Title: Evaluation of [18F]MNI-1126 as an Imaging Marker for Synaptic Density Loss in the Brain of Patients With Probable Alzheimer's Disease, Probable Parkinson's Disease (PD) Subjects as Compared to Healthy Volunteers (HV).
Brief Title: Evaluation of [18F]MNI-1126 as an Imaging Marker for Synaptic Density Loss
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Invicro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: [18F]MNI-1126
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Alzheimer Disease; Parkinson Disease; Healthy Volunteers
Keywords: AD; PD; HV
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]MNI-1126 (Experimental): To measure the dynamic uptake and washout of [18F]MNI-1126 in the brain using positron emission tomography (PET) in subjects with AD, PD, and healthy volunteers.
  Interventions: Drug: [18F]MNI-1126

INTERVENTIONS:
Drug: [18F]MNI-1126 — Florbetapir PET imaging will be completed in all healthy volunteers and AD subjects as part of the screening procedures.
  DaTscan SPECT imaging will be completed in those PDsubjects who have not previously had DaTscan imaging as part of the screening procedures.

SUMMARY:
The primary objective of this protocol is to examine [18F]MNI-1126 as a tool to assess synaptic density loss.

DETAILED DESCRIPTION:
The primary objective of this protocol is to examine [18F]MNI-1126 as a tool to assess synaptic density loss.The specific objectives are:

* Examine [18F]MNI-1126 as a tool to assess synaptic density loss.
* To measure the dynamic uptake and washout of [18F]MNI-1126 in the brain using positron emission tomography (PET) in subjects with AD, PD, and healthy volunteers.
* To measure blood metabolites of [18F]MNI-1126 and perform kinetic modeling to assess its ability to measure synaptic density loss in the brain using the tracer plasma concentration or a reference region as indirect input.
* To acquire safety data following injection of [18F]MNI-1126.

ELIGIBILITY:
Inclusion Criteria (for all subjects)

* Written informed consent must be obtained before any assessment is performed.
* Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year (i.e. 12 consecutive months with no menses without an alternative medical cause) or, if they are of child-bearing potential, must commit to use two methods of contraception, one of which is a barrier method for the duration of the study.
* Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for male subjects for the study duration.
* Male subjects must not donate sperm for the study duration.
* Willing and able to cooperate with study procedures.
* For females, non-child bearing potential or negative urine pregnancy test on day of [18F]MNI-1126 injection.

Inclusion Criteria PD subjects:

* Are males or females ≥ 30 years of age.
* Must have at least two of the following: resting tremor, bradykinesia, rigidity (must have either resting tremor or bradykinesia); OR either asymmetric resting tremor or asymmetric bradykinesia.
* Have Hoehn and Yahr stage ≤3.
* Have a MMSE score ≥ 22.
* PD subjects may be treated with PD symptomatic therapy on a stable dose of medications for a period of at least 30 days prior to the [18F]MNI-1126 PET imaging visit.
* Have screening or prior DaTscan SPECT imaging demonstrating evidence of dopamine transporter deficit based on visual read.

Healthy volunteers inclusion criteria:

* Males and females aged ≥50 years. Healthy with no clinically relevant finding on physical examination at screening and upon reporting for the [18F]MNI-1126 imaging visit.
* No cognitive impairment from neuropsychological battery as judged by the investigator.
* Have screening or prior ( in the last 12 months ) amyloid PET imaging demonstrating no significant amyloid binding based on qualitative (visual read).
* No family history of Alzheimer's disease or neurological disease associated with dementia.
* Have a CDR global score=0.
* Have an MMSE score ≥28.

Inclusion criteria for subjects with a diagnosis of probable Alzheimer's disease (AD):

* Males and females aged 50 to 80 years.
* Have probable Alzheimer's disease dementia, based on the NINCDS/ADRDA and DSM-IV criteria, with mild severity and amnestic presentation.
* Have a CDR score ≥ 0.5 at screening.
* Have a MMSE score ≤ 28.
* Have screening or prior (in the last 12 months) amyloid PET imaging demonstrating amyloid binding based on qualitative analysis (visual read). Amyloid PET imaging results will be shared with participants, and scans may be used by participants for future research use.
* A brain MRI that supports a diagnosis of AD, with no evidence of significant neurologic pathology (see exclusion criteria).
* Medications taken for symptomatic treatment of AD must be maintained on a stable dosage regimen for at least 30 days before screening visit.
* Signed and dated written informed consent obtained from the subject and the subject's legally authorized representative or caregiver (if applicable).

Exclusion Criteria all subjects:

* Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness.
* Subject has received an investigational drug or device within 30 days of screening
* Prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds the effective dose of 50 mSv, which would be above the acceptable annual limit established by the US Federal Guidelines.
* Pregnancy, lactating or breastfeeding.
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Unsuitable veins for repeated venipuncture.
* MRI exclusion criteria include: Findings that may be responsible for the neurologic status of the patient such as significant evidence of cerebrovascular disease (more than two lacunar infarcts, any territorial infarct >1cm3, or deep white matter abnormality corresponding to an overall Fazekas scale of 3 with at least one confluent hyperintense lesion on the FLAIR sequence that is ≥20 mm in any dimension), infectious disease, space-occupying lesions, normal pressure hydrocephalus or any other abnormalities associated with CNS disease.
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.
* Are claustrophobic or otherwise unable to tolerate the imaging procedure

Exclusion criteria for subjects with AD:

• Has received treatment that targeted Aβ or tau within the last 3 months.

Exclusion criteria for subjects PD:

* Ongoing treatment with methylphenidate, modafinil, metoclopramide, alpha methyldopa, reserpine, or amphetamine derivative for subjects requiring DaTscan imaging.
* Subjects may take stable doses of bupropion, however this medication must be held for at least 12 hours prior to DaTscan imaging.
* Subject has known hypersensitivity to iodine or potassium iodide (KI) in the opinion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Regions in the VOI template will be used to quantify the regional tracer uptake and used for comparison of potential uptake differences across the different groups. | 1 year
  Descriptive statistics will be applied to describe the tau deposition by region as measured by [18F]MNI-1126.

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, M.D., Ph. D, Principal Investigator — Invicro
Locations (1):
- Invicro, New Haven, Connecticut, United States

REFERENCES:
- See also: Invicro home page — http://www.invicro.com